CLINICAL TRIAL: NCT06826560
Title: Evaluation of Immunological, Microbiological and Metabolomic Profiles of Patients with Chronic Obstructive Pulmonary Disease in Selected Clinical Phenotypes.
Brief Title: Evaluation of Immunological, Microbiological and Metabolomic Profiles in COPD
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: NCN-NZ5/00694-1
Record Dates: First submitted 2022-05-31; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: COPD; Emphysema; Chronic Bronchitis; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Induced sputum Plasma Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- COPD patients: Inclusion criteria age ⩾ 40 years, written informed history of smoking ⩾ 10 pack-years COPD diagnosis (post- bronchodilator FEV1/FVC < LLN) stable COPD (min. 3 months criteria for the study.
- Smokers without COPD: age ⩾ 40 years, written informed history of smoking ⩾ 10 pack-years FEV1/FVC≥LLN
- Never-smokers: without <1 pack-year, COPD no current smoking (min. 1 year prior the study) FEV1/FVC≥LLN

SUMMARY:
COPD is a significant health problem worldwide. It affects more than 10% of patients over the age of 40. According to the World Health Organization, it is the third most common cause of death among adults in the world, and the number of patients is continuously growing. Hence, all measures aimed at a better understanding of COPD pathogenesis, the course of the disease, and limitations in treatment efficacy seem critically important. Since 2008 our team has provided a substantial output in understanding the pathophysiology of airway inflammation in obstructive lung diseases. In our studies, we systematically evaluated selected cytokines concentrations in different respiratory samples to determine their mutual relations and to determine the role of cytokines in airway inflammation more precisely. However, there is still a large gap in our understanding of COPD. It is hypothesized that in COPD pathogenesis, additional factors, like genetics, autoimmune processes or deviated microbiota are involved. Each of the mentioned factors leads to a different type of immune response with a different effect on the airways. We believe that using more advanced laboratory methods (i.e. metabolomics and airway microbiome analysis) alongside the well-established ones (i.e. cellular and cytokine composition) will allow for an adequate characterization of inflammation.

The study will include 50 COPD subjects and 50 smokers without COPD and 20 control subjects (never smokers) who meet the inclusion and exclusion criteria (Table 1) and give an informed written consent to participate in the study. All study participants will undergo the following procedures: peripheral blood sample collection, chest HRCT imaging (without contrast), lung function assessment (spirometry with a bronchial obstruction reversibility test, bodyplethismography, diffusion lung capacity for carbon monoxide (DLCO), sputum induction with sterile hypertonic saline (NaCl).

ELIGIBILITY:
Inclusion Criteria:

* age ⩾ 40 years,
* written informed history of smoking ⩾ 10 pack-years
* COPD diagnosis (post- bronchodilator FEV1/FVC < LLN)
* stable COPD (min. 3 months)

Exclusion Criteria:

* history of asthma or current lung disease (exception: solitary nodules), respiratory failure
* use of inhaled or oral steroids in the 3 months prior to the study,
* infection of the respiratory tract or exacerbation in the 3 months prior the study
* uncontrolled comorbidities such as: systemic connective tissue diseases, malignancy, uncontrolled cardiovascular diseases, chronic paranasal sinusitis,
* contraindications to sputum induction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each subject visiting the outpatient clinic at our department presenting exertional dyspnoea and/or chronic cough will be screened for eligibility to participate in the study. A control group (never-smokers) will consist of volunteers matched by age and sex to the study group. Inclusion and exclusion criteria are presented in Table 1. Subjects who gave their written informed consent will be divided into three groups (Table 1). The assignment to a specific study group will be based on past medical history, clinical signs and symptoms, and the results of spirometry with a bronchial obstruction reversibility test.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Development of a Risk Calculator for COPD Severity and Phenotyping Using Feature Selection and Enrichment Analysis | Up to 6 months after sample collection
  In this study, we will use the Boruta algorithm for feature selection and perform enrichment analysis to identify overrepresented biological pathways. Based on these results, we will develop and validate a calculator that generates a risk score for the disease and predicts the likelihood of severe progression. This calculator will serve as an outcome measure, providing an integrated tool to assess patient status and guide clinical decisions.

SECONDARY OUTCOMES:
Secondary Outcome Measure 1: Identification of Omics Biomarkers Associated with CT Imaging Changes in COPD | Up to 6 months after sample collection
  We will apply the Boruta algorithm to proteomic, metabolomic, and cytokine data to identify molecules significantly associated with CT imaging findings (e.g., wall thickening and emphysema). Additionally, we will explore the relationships between inflammatory cytokines, specific metabolites, proteins, and immune cell populations (assessed in induced sputum) to elucidate mechanistic links between systemic inflammation and structural lung alterations.
Secondary Outcome Measure 2: Assessment of Host-Environment Interactions via Microbiome Analysis | Up to 6 months after sample collection
  We will perform microbiome profiling of the airway and integrate these data with proteomic, metabolomic, cytokine, and immune cell information from induced sputum using the Boruta algorithm. This analysis will assess host-environment interactions by identifying biomarkers that connect microbial composition with inflammatory profiles and CT imaging changes, thereby enhancing our understanding of the interplay between host factors and environmental influences in COPD.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Banacha Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No